CLINICAL TRIAL: NCT06017258
Title: Phase I Trial of CLEc12a (CD371) Targeted ArmoRed Immune Effector Cells in Patients With Relapsed/Refractory Acute Myeloid Leukemia (CLEAR-AML)
Brief Title: A Study of CD371-YSNVZIL-18 CAR T Cells in People With Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-016
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Refractory Acute Myeloid Leukemia; Relapsed Acute Myeloid Leukemia; Acute Myeloid Leukemia; Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory
Keywords: Refractory Acute Myeloid Leukemia; Relapsed Acute Myeloid Leukemia; Acute Myeloid Leukemia; Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory; ArmoRed; CLEAR-AML; CLEc12a; CD371; Memorial Sloan Kettering Cancer Center; 23-016
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1 (Experimental): Participants with Relapsed/Refractory Acute Myeloid Leukemia (R/R AML)
  Interventions: Biological: CD371-specific/YSNVz/I-18 CAR T cells
- Dose Level 2 (Experimental): Participants with Relapsed/Refractory Acute Myeloid Leukemia (R/R AML)
  Interventions: Biological: CD371-specific/YSNVz/I-18 CAR T cells
- Step-Down Dose (Experimental): Participants with Relapsed/Refractory Acute Myeloid Leukemia (R/R AML)
  Interventions: Biological: CD371-specific/YSNVz/I-18 CAR T cells

INTERVENTIONS:
Biological: CD371-specific/YSNVz/I-18 CAR T cells — Cohorts will be infused with escalating doses of CD371-specific/YSNVz/IL-18 CAR T cells with lymphodepleting chemotherapy (LDC) to establish the maximum tolerated dose (MTD). There is a third, lower dose level (step-down dose) available for dose de-escalation in the event of severe toxicity at the first planned dose level.

SUMMARY:
The purpose of this study is to find out whether CD371-YSNVZ-IL18 CAR T cells are safe, and to look for the highest dose of CD371-YSNVZ-IL18 CAR T cells that cause few or mild side effects in participants.

ELIGIBILITY:
Inclusion Criteria:

Subject Inclusion: Collection of T cells (Part A)

* History of CD371+ AML

  * Any disease status is eligible for collection
  * Expression of CD371 at any level on AML blasts (any method of detection including IHC and/or flow cytometry)
* Age/Weight

  * Pediatrics: ≥ 1 year and ≥ 10kg for collection
  * Adults: no limit on age/weight for collection
* Patients with history of allo-HCT are eligible for collection if:

  * ≥ 100 days post-transplant
  * no evidence of active GVHD
  * off any immunosuppressive agents for 30 days prior to collection (physiologic dose of corticosteroids is acceptable)

Subject Inclusion: Treatment with CD371-specific/YSNVz/IL-18 CAR T cells (Part B)

* Relapsed/Refractory CD371+ AML (meeting criteria defined below) for primary refractory AML, late first relapse, and/or advanced disease:

  o Primary refractory AML: Patients are eligible from disease perspective in the event of failure to achieve a CR, CRh or CRi after one or more of the following regimens:
* Two or more courses of standard intensive induction chemotherapy (e.g., cytarabine and daunorubicin given as "7+3," MEC, HiDAC, FLAG+idarubicin, etc.);
* Two or more cycles of venetoclax in combination with one of the following (azacitidine OR decitabine OR low-dose cytarabine), with or without other agents;
* Six or more cycles of azacitidine monotherapy OR four or more courses of decitabine monotherapy

  * Early first relapse: Patients are eligible from disease perspective in the event of first morphologic relapse or new extramedullary disease less than 12 months after previously having achieved CR, CRh, or CRi following AML-directed therapy
  * Late first relapse: Patients with first morphologic relapse or new extramedullary disease ≥12 months after previously having achieved CR, CRh, or CRi following AML-directed therapy may respond to intensive re-induction using the initial induction regimen and not eligible from a disease perspective unless the treating investigator feels the patient is unlikely to benefit from repeating the initial induction regimen (for example, relapse occurring 12 months into CR on continuous azacitidine/venetoclax therapy), in which case the rationale for considering enrollment must be clearly documented and risks, benefits, and alternatives discussed with the patient.
  * Advanced disease: Patients are eligible from disease perspective in the event of relapsed AML refractory to reinduction therapy, relapse following alloHCT, or second or later relapse.
  * Disease eligibility considerations for all patients: Patients with relapsed or refractory AML with susceptible mutations for which there is an FDA approved therapy (for example, IDH1 mutation, ivosidenib; IDH2 mutation, enasidenib; FLT3-ITD/TKD, gilteritinib) are not eligible from a disease perspective unless they meet one or more of the below criteria:
* Failure to achieve CR, CRh, or CRi following therapy with one or more targeted therapies for relapsed or refractory AML directed to the actionable mutation(s);
* Intolerance of one or more targeted therapies for relapsed or refractory AML directed to the actionable mutation(s);
* Treating investigator feels the patient would be unlikely to benefit from FDA-approved targeted therapy based on disease characteristics, in which case the rationale for considering enrollment must be clearly documented and risks, benefits, and alternatives discussed with the patient Age: any age is eligible for treatment if eligible for collection

  o The first 3 patients in the first dose cohort must be ≥ 16 years of age, while the first 2 patients in subsequent cohorts must be ≥ 16 years of age (see Section 10.4)
* Adequate performance status:

  * Age ≥ 16 years: ECOG ≤ 1 or Karnosfsky ≥ 60
  * Age < 16 years: Lansky ≥ 60
* Patients with history of allo-HCT are eligible for treatment if:

  * ≥ 100 days post-transplant
  * no evidence of active GVHD
  * off any systemic immunosuppressive agents for 30 days prior to treatment (physiologic dose of corticosteroids is acceptable)
  * Treating physician considers the patient to be a candidate for second alloHCT
* Identification of a suitable donor/source for alloHCT as determined by the treating physician.
* Adequate organ function is required, defined as follows:

  * Hepatic: Serum total bilirubin ≤ 1.5 mg/dL, unless benign congenital hyperbilirubinemia or unless thought to be disease related.
  * Hepatic: ALT and AST < 3 times the upper limit of normal unless thought to be disease-related.
  * Renal: serum creatinine < 2.0 mg/100 ml (> 18 years) or ≤ 2.5 x institutional upper limit of normal (ULN) for age
* If serum creatinine is outside the normal range, then CrCl > 40 mL/min/1.73m2 (calculated or estimated) or GFR (mL/min/1.73m2) > 40% of predicted normal for age.

Normal GFR by Age Age: 1 week / Mean GFR +/-SD (mL/min/1.73 m2): 40.6 + / - 14.8 Age: 2 - 8 weeks / Mean GFR +/-SD (mL/min/1.73 m2): 65.8 + / - 24.8 Age: > 8 weeks / Mean GFR +/-SD (mL/min/1.73 m2): 95.7 +/- 21.7 Age: 2 - 12 years / Mean GFR +/-SD (mL/min/1.73 m2): 133 +/- 27 Age: 13 - 21 years (males) / Mean GFR +/-SD (mL/min/1.73 m2): 140 +/- 30 Age: 13 - 21 years (females) / Mean GFR +/-SD (mL/min/1.73 m2): 126.0 + / - 22.0 Abbreviations: GFR, glomerular f filtration rate; SD, standard deviation

* Greater than 2 years old: Normal GFR is 100 mL/min/1.73m2.
* Infants: GFR must be corrected for body surface area.

  * Cardiac: LVEF ≥ 50% by MUGA or resting echocardiogram.
  * Pulmonary: Adequate pulmonary function as assessed by ≥ 92% oxygen saturation on room air by pulse oximetry

Exclusion Criteria:

Subject Exclusion: Collection of T cells (Part A)

* Pregnant or lactating women; women of childbearing age, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception while receiving study treatment and for at least 12 months after all treatment is finished
* Sexually active males, unless they are willing to use a condom during intercourse while receiving study treatment and for at least 12 months after all treatment is finished
* Radiographically-detected or symptomatic CNS disease or CNS 3 disease (i.e., presence of ≥ 5/ul WBC in CSF). Subjects with adequately treated CNS leukemia are eligible.
* Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject
* Impaired cardiac function (LVEF < 50%) as assessed by ECHO or MUGA scan
* Patients with following cardiac conditions will be excluded:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure
  * Myocardial infarction ≤ 6 months prior to enrollment
  * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
* Positive serologic test results for HIV
* Acute or chronic HBV infection as assessed by serologic (HBVsAg) or PCR results, defined as HBVsAg+, HBVcAb+, HBV PCR+.
* Acute or chronic HCV infection as assessed by serologic (HCV ab) or PCR results, defined as HCV Ab+ with reflex to positive HCV PCR
* Patient/parent/LAR unable to give informed consent/

Subject Exclusion: Treatment with CD371-specific/YSNVz/IL-18 CAR T cells (Part B)

* Bridging chemotherapy occurring < 1 week prior to administration of LDC

  o Exception: hydroxyurea can be continued up to 72 hours prior to leukapheresis or 24 hours prior to LDC
* Pregnant or lactating women
* Radiographically-detected or symptomatic CNS disease or CNS 3 disease (i.e., presence of ≥ 5/ul WBC in CSF). Subjects with adequately treated CNS leukemia are eligible.
* Isolated extramedullary disease
* Lack of a suitable donor/source for allogeneic HSCT as determined by the treating physician.
* Patients with prior alloHCT are allowed as long as alloHCT occurred ≥100 days prior to date of treatment with CD371-specific/YSNVz/IL-18 CAR T cells and as long as the patient is without ongoing requirement for systemic graft-versus-host therapy
* Uncontrolled, symptomatic, intercurrent illness including but not limited to infection, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject
* Impaired cardiac function (LVEF < 50%) as assessed by ECHO or MUGA scan.
* Patients with following cardiac conditions will be excluded:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure
  * Myocardial infarction ≤ 6 months prior to enrollment
  * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
* Positive serologic test results for HIV.
* Acute or chronic HBV infection as assessed by serologic (HBVsAg) or PCR results, defined as HBVsAg+, HBVcAb+, HBV PCR+.
* Acute or chronic HCV infection as assessed by serologic (HCV ab) or PCR results, defined as HCV Ab+ with reflex to positive HCV PCR
* Active second malignancy that requires systemic treatments, with the exception of malignancy treated with curative intent and without evidence of disease for > 2 years before screening
* Patient/parent/LAR unable to give informed consent
* Any other condition/issue which, in the opinion of the treating physician, would make the patient ineligible for the study; conditions that in the Principal Investigator's opinion might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2026-08-22 (Estimated); Study Completion 2026-08-22 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of CAR T cells | up to 6 months
  Determine the Maximum Tolerated Dose/MTD of CAR T cells in participants with Relapsed/Refractory Acute Myeloid Leukemia (R/R AML)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Geyer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Geyer MB, DeWolf S, Mi X, Weis K, Shaffer BC, Cadzin B, McAvoy D, Katsamakis Z, Lorenc R, Lewis AM, Gipson B, Cuibus MA, Girotra NN, Wu K, Smith N, Burns ER, Um JS, Yoo S, Masouleh BK, Galera P, Hosszu K, Chaudhari J, Wang X, Lin Q, Curran KJ, Park JH, Scheinberg DA, van den Brink MRM, Abdel-Wahab O, Brentjens RJ, Daniyan AF. CD371-targeted CAR T cells secreting interleukin-18 exhibit robust expansion and clear refractory acute myeloid leukemia. Blood. 2025 Dec 25;146(26):3163-3174. doi: 10.1182/blood.2025029532. PMID 40864984
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org